CLINICAL TRIAL: NCT00297830
Title: Zoledronic Acid Versus Alendronate for Prevention of Bone Loss After Organ Transplantation
Acronym: CTX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Elizabeth Shane, Professor of Medicine, Endocrinology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAB2324; CZOL446H104 (Other: Novartis)
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Heart Transplantation; Liver Transplantation; Bone Resorption
Keywords: Heart Transplantation; Liver Transplantation; Immunosuppression; Bone Density/drug effects; Alendronate; Zoledronic acid; Comparative study; Humans
MeSH Terms: conditions — Bone Resorption | interventions — Zoledronic Acid; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Zoledronic Acid & Placebo Alendronate (Experimental): Group 1 will receive an infusion of active zoledronic acid 5 mg during the first 4 weeks after transplantation. Placebo alendronate 70 mg once weekly will be initiated at the same time as the first zoledronic acid infusion.
  Interventions: Drug: Zoledronic acid; Other: Placebo Alendronate
- Placebo Zoledronic Acid & Active Alendronate (Experimental): Group 2 will receive an infusion of placebo zoledronic acid during the first 5 weeks after transplantation. Active alendronate 70 mg once weekly will be initiated at the same time as the placebo infusion.
  Interventions: Drug: Alendronate; Other: Placebo Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid — Drug is administered through 5 mg intravenous infusion over 20 minutes
  Other Names: Zometa
  Arms: Active Zoledronic Acid & Placebo Alendronate
Drug: Alendronate — Alendronate 70 mg will be taken once a week in the morning at least 30-60 minutes before first meal
  Other Names: Fosamax
  Arms: Placebo Zoledronic Acid & Active Alendronate
Other: Placebo Zoledronic Acid — Infusion of placebo zoledronic acid during the first 5 weeks after transplantation
  Arms: Placebo Zoledronic Acid & Active Alendronate
Other: Placebo Alendronate — Placebo alendronate 70 mg once weekly
  Arms: Active Zoledronic Acid & Placebo Alendronate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of zoledronic acid with alendronate in the prevention of bone loss after organ transplantation. Zoledronic acid is given as a single intravenous infusion. Alendronate is given as a weekly pill. Both are expected to be very effective, but it is not known which one will work best.

DETAILED DESCRIPTION:
Patients who have undergone heart or liver transplantation are usually required to remain on medications, such as Prednisone and Cyclosporine A or Tacrolimus, that prevent the body from rejecting the transplanted organ. These medications may cause bone loss which leads to thinning of the bones (osteoporosis) and therefore greatly increase the risk of having broken bones (fractures) after transplantation. Several published studies have shown that 14% to 35% of heart transplant patients develop fractures (spine, ribs and hip) during the first year after transplantation. We have previously shown that alendronate (Fosamax), a drug approved by the FDA for prevention and treatment of postmenopausal osteoporosis and prednisone-induced osteoporosis, prevents bone loss after heart transplantation. We are conducting this study to determine whether a newer drug, zoledronic acid, is as effective as alendronate.

This study is a randomized, double-blind, placebo-controlled 2-year study. Participants will receive one dose of active zoledronic acid during the first month after heart or liver transplantation and weekly placebo alendronate pills or one dose of placebo zoledronic acid and weekly active alendronate pills for the first year after transplant. Over 2 years, participants will provide blood samples on nine occasions. Bone density will be performed 4-5 times and spine xrays will be performed twice.

ELIGIBILITY:
Inclusion Criteria:

* A man or woman, aged 20 to 70, of any race who has had a heart or liver transplant

Exclusion Criteria:

* hyperparathyroidism
* Paget's disease
* hyperthyroidism
* cancer
* severe kidney disease,
* intestinal disease
* active peptic ulcer disease
* current or past treatment for osteoporosis
* pregnancy or lactation
* severe oral/dental disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shane E, Addesso V, Namerow PB, McMahon DJ, Lo SH, Staron RB, Zucker M, Pardi S, Maybaum S, Mancini D. Alendronate versus calcitriol for the prevention of bone loss after cardiac transplantation. N Engl J Med. 2004 Feb 19;350(8):767-76. doi: 10.1056/NEJMoa035617. PMID 14973216
- [Result] Shane E, Cohen A, Stein EM, McMahon DJ, Zhang C, Young P, Pandit K, Staron RB, Verna EC, Brown R, Restaino S, Mancini D. Zoledronic acid versus alendronate for the prevention of bone loss after heart or liver transplantation. J Clin Endocrinol Metab. 2012 Dec;97(12):4481-90. doi: 10.1210/jc.2012-2804. Epub 2012 Sep 28. PMID 23024190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women, aged 20 to 70 yr, who had undergone heart or liver transplantation at CUMC were eligible. Of 495 patients transplanted between 3/2006 and 7/2009, 235 were ineligible. 149 patients declined or were not approached. 84 were randomized, 43 to alendronate and 41 to zoledronate. 27 were the reference group since they refused randomization.
Pre-assignment Details: Serum creatinine levels above 2.0 mg/dl, or enrollment in another clinical trial
Groups:
- Active Zoledronic Acid and Placebo Alendronate: Group 1 will receive an infusion of active zoledronic acid 5 mg during the first 4 weeks after transplantation. Placebo alendronate 70 mg once weekly will be initiated at the same time as the first zoledronic acid infusion.
- Placebo Zoledronic Acid and Active Alendronate: Group 2 will receive an infusion of placebo during the first 5 weeks after transplantation. Active alendronate 70 mg once weekly will be initiated at the same time as the placebo infusion.
- Reference Group: The reference group included concurrently transplanted patients with T scores of -1.5 or greater.
Period: Baseline
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Started | 41 | 43 | 27
Completed | 41 | 43 | 27
Not Completed | 0 | 0 | 0
Period: 6 Month Visit
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Started | 41 | 43 | 27
Completed | 38 | 41 | 24
Not Completed | 3 | 2 | 3
Not completed — Death | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0
Period: 12 Month Visit
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Started | 38 | 41 | 24
Completed | 37 | 35 | 24
Not Completed | 1 | 6 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Based on preliminary data that total hip BMD would decrease by 1.5 ± 3.7% on alendronate and increase by 1.0 ± 3.7% on zoledronate, we estimated that 35 subjects per group would provide 80% power and 5% α to detect a 2.5 ± 3.7% difference between randomized groups. Anticipating a 20% dropout, 84 subjects were randomized.
Groups:
- Placebo Infusion and Active Alendronate: Group 2 will receive an infusion of placebo during the first 5 weeks after transplantation. Active alendronate 70 mg once weekly will be initiated at the same time as the placebo infusion.
- Total: Total of all reporting groups
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Infusion and Active Alendronate | Reference Group | Total
Number analyzed (Participants) | 41 | 43 | 27 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8) | 54 (10) | 48 (15) | 52.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 7 | 26
  Male | 30 | 35 | 20 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 12 | 5 | 21
  Not Hispanic or Latino | 37 | 31 | 22 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Total Hip Bone Mineral Density (BMD) at 12 Months
Description: BMD was measured by dual-energy x-ray absorptiometry (QDR-4500 densitometer; Hologic, Inc., Bedford, MA); short-term in vivo coefficient of variation is 0.68% (spine) and 1.36% (femoral neck). T scores were generated using gender-specific databases provided by the manufacturer.
Time Frame: Baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Number analyzed (Participants) | 37 | 35 | 24
percent change | 0.39 [-0.64 to 1.42] | -0.21 [-1.25 to 0.84] | -2.2 [-3.6 to -0.7]

2. Secondary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 12 Months
Description: as for outcome 1
Time Frame: Baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Number analyzed (Participants) | 37 | 35 | 24
percent change | 1.98 [0.55 to 3.40] | -0.45 [-1.88 to 0.99] | -2.6 [-4.4 to -0.9]

3. Secondary Outcome: Percentage Change From Baseline in Femoral Neck Bone Mineral Density (BMD) at 12 Months
Description: as for outcome 1
Time Frame: Baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Number analyzed (Participants) | 37 | 35 | 24
percent change | 0.28 [-1.16 to 1.71] | -0.57 [-2.02 to 0.88] | -3.3 [-4.8 to -1.8]

4. Secondary Outcome: Serum N-telopeplide Percent Change
Time Frame: 24 months
Population: Serum n-telopeplide percent change was not collected.
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Zoledronic Acid and Active Alendronate | Reference Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo Infusion and Active Alendronate: Group 2 will receive an infusion of placebo during the first 5 weeks after transplantation. Active alendronate 70 mg once weekly will be initiated at the same time as the placebo infusion.https://register.clinicaltrials.gov/prs/html/results_definitions.html#Result_ParticipantFlow_Period_title
Arm/Group | Active Zoledronic Acid and Placebo Alendronate | Placebo Infusion and Active Alendronate | Reference Group
Serious Adverse Events (participants affected / at risk) | 21/41 | 14/43 | 2/27
Other Adverse Events (participants affected / at risk) | 14/41 | 11/43 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Zoledronic Acid and Placebo Alendronate (N=41) | Placebo Infusion and Active Alendronate (N=43) | Reference Group (N=27)
Death (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hospitalization (General disorders) | 20 (20) | 14 (14) | 0 (0) — Includes all hospital readmissions after randomization or enrollment.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Zoledronic Acid and Placebo Alendronate (N=41) | Placebo Infusion and Active Alendronate (N=43) | Reference Group (N=27)
Infection (Infections and infestations) | 14 (14) | 11 (11) | 0 (0) — Includes all infections due to cytomegalovirus and all other infections that necessitated hospitalization, intravenous antibiotic therapy, or both.
Rejection (General disorders) | 4 (4) | 2 (2) | 0 (0) — Rejection after month 1 necessitating change in immunosuppressive regimen
Flu-like symptoms after zoledronate or matching placebo (General disorders) | 2 (2) | 1 (1) | 0 (0)
Hypocalcemia (Endocrine disorders) | 4 (4) | 5 (5) | 0 (0) — Albumin-corrected serum calcium below 8.0 mg/dL. To convert values for serum calcium to millimoles per liter, multiply by 0.2495.
Serum Calcium > 2.0 mg/dL (Endocrine disorders) | 1 (1) | 7 (7) | 0 (0) — At any visit after randomization. To convert values for serum creatinine to millimoles per liter, multiply by 88.4.
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Heart and liver transplant recipients differ in pretransplant bone disease and exposure to prednisone. Not powered to detect differences in fracture rates,an important clinical outcome,one that would require a large comparative effectiveness trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No